CLINICAL TRIAL: NCT00309309
Title: A Prospective, Longitudinal Study to Assess the Metabolic and Renal Effects of Rosiglitazone in Albuminuric Kidney Transplant Recipients
Brief Title: Metabolic and Renal Effects of Rosiglitazone in Kidney Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLITA-TX
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone

SUMMARY:
Abnormalities in glucidic and lipidic metabolism are common features in renal transplant patients on chronic immunossupression with steroids and calcineurin inhibitors. In kidney transplant patients with chronic rejection these abnormalities cluster with renal and cardiovascular risk factors and altogether may sustain premature graft loss and may increase the risk of cardiovascular morbidity and mortality. Thiozolidinediones are a new class of oral antidiabetic agents that may increase insulin sensitivity improving the glucose tolerance and dyslipidemia. Moreover, rosiglitazone -one of these drugs- has been reported to decrease blood pressure and albuminuria in subjects with type 2 diabetes and nephropathy. Recent finding that glitazones ameliorate the glucidic and lipidic profile induced by steroid treatment in healthy subjects, provided a further rationale to evaluate the metabolic and renal effects of glitazones in renal transplant patients on chronic steroid therapy. Thus, we designed and organized a pilot study to assess the short-term risk/benefit profile of rosiglitazone in renal transplant patients with chronic rejection. Ten patients will have a basal evaluation of insulin sensitivity, glucose tolerance,lipid profile, renal hemodynamic and albuminuria. These evaluations will be repeated at the end of the treatment (4 months of therapy with rosiglitazone 8 mg/day) period and 2 months after treatment withdrawal.

DETAILED DESCRIPTION:
INTRODUCTION Decreased insulin sensitivity, impaired glucose tolerance and dyslipidemia are common features in renal transplant patients on chronic immunosuppression with steroids and calcineurine inhibitors. In renal transplant patients with chronic allograft dysfunction these metabolic abnormalities typically cluster with well-established renal and cardiovascular risk-factors such as hypertension and albuminuria. Altogether these factors may sustain and accelerate the progression of chronic allograft dysfunction to end stage renal disease (ESRD) and increase the risk of premature cardiovascular morbidity and mortality.

Thiazolidinediones (glitazones) are a new class of oral antidiabetic agents that may increase insulin sensitivity through activation of the peroxisome prolipherator-activated receptor gamma (PPARgamma). By ameliorating insulin sensitivity, these drugs may also improve glucose tolerance and dyslipidemia. These properties have led to their current utility as antidiabetic drugs. Moreover, finding that one of these drugs - rosiglitazone - has been reported to decrease arterial blood pressure and albuminuria in patients with type 2 diabetes and nephropathy, has been taken to suggest that glitazones may also have a specific reno- and cardio-protective effect. This effect could specifically apply to renal transplant patients with chronic allograft dysfunction in whom glitazones, in addition to ameliorate insulin resistance, glucose tolerance and dyslipidemia, might help controlling arterial hypertension and reducing albuminuria.

Recent finding that glitazones ameliorate the insulin resistant status induced by steroid treatment in healthy subjects, provides a further rationale to evaluate the metabolic and renal effects of glitazones in renal transplant patients on chronic steroid therapy.

AIM To evaluate the short-term risk/benefit profile of rosiglitazone treatment in renal transplant patients with chronic allograft dysfunction.

DESIGN After a basal evaluation of systolic/diastolic blood pressure,body weight, insulin sensitivity (by euglycemic hyperinsulinemic clamp), glucose tolerance (by standard glucose tolerance test), lipid profile, renal hemodynamics (GFR and RPF by inulin and PAH renal clearances, respectively), albuminuria (mean of three consecutive overnight urine collections), albumin, IgG, Na+ and free water fractional clearances and other routine laboratory analyses, patients satisfying the selection criteria will enter 4-month therapy with rosiglitazone 4 mg/day, up-titrated, if well-tolerated, to 8 mg/day 4 weeks later. Baseline evaluations will be repeated at the end of the treatment period and 2 months after treatment withdrawal. Blood pressure, body weight and routine laboratory tests - including liver function tests - will be evaluated also at 1 and 2 weeks of rosiglitazone therapy, at month 1 and then every month up to study end. Albuminuria will also be evaluated at month 2 of rosiglitazone therapy.

No major change in diet and immunosuppressive, antihypertensive and other concomitant treatments will be introduced throughout the whole study period. A low salt (2 grams of Na+ per day) and a controlled dietary protein intake (0.8 g/kg/body weight per day) will be recommended to all patients. Should any evidence of clinically relevant water retention or of liver toxicity occur throughout the treatment period, rosiglitazone will be back-titrated to the initial dose or withdrawn as deemed clinically appropriate.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-70 years old
* kidney transplant since at least six months
* serum creatinine ≤ 3mg/dl without dialysis requirement
* serum creatinine changes ≤ + 30 % over the last three months
* overnight urinary albumin excretion rate ≥20µg/min
* well controlled hypertension (systolic/diastolic blood pressure <150/90 mmHg)
* concomitant treatment with inhibitors of the renin angiotensin system (RAS) since at least six months
* effective contraception
* written informed consent
* legal capacity

Exclusion Criteria:

* acute graft rejection over the last six months
* immunosuppressive therapy with FK506
* evidence of previous or concomitant liver disease and abnormal liver transaminases over the last six months
* evidence of heart failure (NYHA class II or more) or fluid overload
* overt diabetes or concomitant treatment with oral antidiabetic agents and/or insulin
* specific contraindication to the study drug
* legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (at 0,4,6 months)
Blood pressure (at 0,4,6 months)
Albumin urinary excretion (at 0,4,6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Perico, MD, Principal Investigator — Mario Negri Institute
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy